CLINICAL TRIAL: NCT06594419
Title: Efficacy of the Healthy Mother Healthy Baby Toolkit for Maternal and Child Nutrition in Ethiopia
Brief Title: Healthy Baby Healthy Mother Toolkit
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Agency Fund and GDI solutions, LLC (Unknown); Amharic Public Health Institute (APHI) (Unknown)
Responsible Party: Principal Investigator, Amy Webb Girard, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00006236
Record Dates: First submitted 2024-08-27; First posted 2024-09-19 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Maternal Nutrition; Child Nutrition
Keywords: Healthy Mother Healthy Baby Toolkit; Maternal nutrition; Health Belief Model
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy Mother Healthy Baby Toolkit (Experimental): 297 women will be enrolled in this arm.
  Interventions: Behavioral: Healthy Mother Healthy Baby Toolkit
- Standard of Care (Active Comparator): 297 women will be enrolled in this arm.
  Interventions: Other: Standard of care

INTERVENTIONS:
Behavioral: Healthy Mother Healthy Baby Toolkit — Customized bowl with markings to indicate the recommended amount of food that participants should consume in pregnancy and while exclusively breastfeeding in the first 6 months, as well as how much they should feed their babies at 6-8 months, 9-12 months, and 1-2 years respectively. The toolkit also includes a spoon used to test and ensure adequate thickness of the meals fed to infants >6mos and a counseling card that indicates the frequency of meals, recommended food groups for meeting daily nutrient needs, and hand hygiene and hygienic food preparation
  Arms: Healthy Mother Healthy Baby Toolkit
Other: Standard of care — The Ethiopian government and Saving Little Lives Initiative (SLL) standard of care includes maternal and infant nutrition education and counseling, iron and folic acid supplementation, as well as training on effective Kangaroo Mother Care (KMC), primarily defined as exclusive breastfeeding and skin-to-skin contact ≥ 8 hours per day-in the event of Low birth weight (LBW) or preterm delivery.
  Arms: Standard of Care

SUMMARY:
The objective of the research is to test whether integrating a mother-baby nutrition toolkit into routine antenatal care service can improve maternal and infant nutrition in Amhara, Ethiopia

DETAILED DESCRIPTION:
The high burden of undernutrition through the critical first 1,000 days persists in Ethiopia. Studies have indicated that approximately 1 in 4 women of reproductive age in Ethiopia are underweight, 17% of babies are born at low birth weight and nearly 50% of children are stunted by age 2. Inadequate diets of pregnant and breastfeeding women, both suboptimal quality and quantity, are a key contributor to maternal and infant undernutrition in Ethiopia.

The National Nutrition Strategy of Ethiopia, adopted in 2008, recommends one additional meal per day to support healthy pregnancy, and two extra meals per day to support lactation (US Agency for International Development (USAID), 2008).

Using the Health Belief Model for behavior change, the study team developed and has tested in other contexts a Healthy Baby Toolkit (HBT) designed to serve as a cue to action to improve maternal and family self-efficacy in providing mothers and their babies with adequate nutrition. The toolkit has previously been tested in India, Kenya, Malawi, and Ethiopia where it has demonstrated acceptability and feasibility, and demonstrated improvement in the diets of children between 6-23 months. This new trial aims to understand the added health benefits of introducing the toolkit to mothers during pregnancy and the early postpartum period when crucial child growth and development trajectories are established.

The study will evaluate the benefits of HBT on maternal nutrition and infant growth, especially during the first 500 days (pregnancy and first 6 months of life). It will also assess strategies for facility and community-based delivery of the toolkit for future rollout and scaling up. Findings from this study will create an evidence base for effective counseling strategies and support advocacy efforts to integrate the toolkit into routine nutrition education and counseling programs in Ethiopia.

ELIGIBILITY:
Inclusion Criteria:

* <20 weeks gestation as determined by maternal report of last menstrual period
* Intending to breastfeed and provide age-appropriate complementary feeding
* Intend to continue services at the health center where they enrolled until their infant is at least 10 months old

Exclusion Criteria:

* Women who participated in the formative phase of the HMHBT project
* Women with an existing medical condition that merits precautions for a high-risk pregnancy and may affect study outcomes independently of the intervention. These include for example, uncontrolled or advanced diabetes, advanced kidney disease (stage 3 or higher); thyroid disease, autoimmune disorders such as lupus, moderate to severe rheumatoid arthritis, organ transplant; blood clotting or bleeding disorders, multiple sclerosis.
* Women with a history of previous preterm delivery (<32w) or very low birth weight babies (<1.5kg)
* Known history of serious obstetric complications that place the mother at increased risk for subsequent adverse events or complications. These include for example multiple miscarriages or stillbirths (>2); eclampsia, hemorrhage, placenta previa, placental abruption, uterine rupture
* Women experiencing pregnancy loss, and neonatal or infant mortality will be excluded from further follow-up. Women who give birth to multiples will be retained but their data will be analyzed separately

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 594 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Maternal Weight gain during pregnancy | Baseline, third trimester
  Maternal weight is measured using a high quality electronic scale (precision 0.10 kg)- SECA (UNICEF).
Infant Birth Weight | At the time of birth
  Infant birthweight will be collected as soon as possible after birth and at most within one week of birth. Birth weight captured by nurses immediately after delivery will be collected from health registers if the mother delivers in the facility, from the Antenatal care (ANC) card or by Research Assistants (RA) if she delivers at home

SECONDARY OUTCOMES:
Infant Weight for age z scores | 7 days post birth, 4 months post birth, 9 months post birth
  Naked or near naked weight is measured using a SECA taring, mother baby scale accurate to 10 g. Readings are made to the nearest 10 g.
  Weight and age in months will be used to estimate weight for age z scores following WHO guidelines.
Infant Length for age Z scores | 7 days post birth, 4 months post birth, 9 months post birth
  Recumbent length is measured using a wooden Schorr measuring board by two trained researchers. One applies gentle traction to bring the crown of the child's head into contact with the fixed headboard; the second holds the baby's feet, without shoes and with toes pointing directly upward, and keeping the knees straight, brings the movable footboard to rest firmly against the heels.
  Length and age in months will be used to estimate length for age z scores following WHO guidelines.
Infant Weight for Length Z scores | 7 days post birth, 4 months post birth, 9 months post birth
  Infant weight and length will be used to estimate z scores following WHO guidelines
Maternal Anthropometry: Mid-upper arm circumference | Baseline, Late pregnancy (32-42 weeks of gestation), 4 months, 9 months postpartum
  Women's mid-upper-arm circumference (MUAC) is measured at enrollment and again at every follow-up period delivery. MUAC is measured using a flexible, non-stretchable tape at the mid-point of the non dominant upper arm, between the acromion process and the tip of the olecranon. The measurement is taken to the nearest mm.
Maternal Anthropometry: Height | Baseline
  A standardized stadiometer is employed, ensuring precision to the nearest 0.1 cm. Women are measured without shoes, wearing light clothing, and with the spine erect and heels together. The measurement is taken from the crown of the head to the bottom of the feet.
Maternal Dietary Data | Baseline, Third trimester, 4 months post partum, 9 months postpartum
  Energy (Kcal/ day) and protein intakes and dietary patterns of participating women will be assessed using a food frequency questionnaire that queries the frequency of consumption and portion size of approximately 80-120 foods over the previous 30 days.
  The 24hr recall will utilize food scales, common utensils (e.g., traditional spoons and bowls, the Healthy Mother Healthy Baby Toolkit (HMHBT) cups), food pictures, and standardized recipes to assist in estimating food amounts (in grams) consumed by pregnant / breastfeeding women
Women's dietary diversity scores | Baseline, third trimester, 4 months post partum and 9 months post partum
  Percentage of women meeting minimum dietary diversity from enrollment through 9month postpartum
Minimum acceptable diet | within 1 week of delivery, 4 months post birth, 9 months post birth
  Summary indicator of infant diet quality assessed at 9 months of age using WHO-approved and validated indicators following a 24-hour recall approach. This outcome is an aggregate indicator comprised of three separate indicators including meeting minimum dietary diversity, minimum meal frequency, and age-appropriate breastfeeding
Exclusive breastfeeding | 1 week postpartum, 4 months postpartum
  A WHO-approved and validated survey tool will be used based on a 24-hour recall of fluids and food intake.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Webb Girard, PhD BSN, Principal Investigator — Rollins School of Public Health
Locations (2):
- Ethiopia (2):
  - Emory University in Ethiopia, Bahir Dar, Amhara
  - Bahir Dar City Zone Health Department, Bahir Dar, Woreda